CLINICAL TRIAL: NCT05792800
Title: Dental Practitioners' Knowledge, Attitudes, and Practice (KAP) Regarding Caries Preventive Measures in Cairo Compared to Riyadh: A Cross-Sectional Study
Brief Title: Dental Practitioners KAP Regarding Caries Preventive Measures in Cairo and Riyadah
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdulmajeed Fahad Mohammed Albishri, Principal Investigator, Cairo University
Other Study IDs: KAP Caries Preventive Measures
Record Dates: First submitted 2023-03-19; First posted 2023-03-31 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Tooth Diseases; Caries,Dental
MeSH Terms: conditions — Tooth Diseases; Dental Caries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to evaluate the knowledge, attitude, and practice of dental practitioners from Cairo and Riyadh regarding caries preventive measures.

DETAILED DESCRIPTION:
Periodontal disease and dental caries have been regarded as the two most enormous worldwide health burdens. Currently, the distribution and severity fluctuate within a single nation or area and throughout the globe. According to epidemiological statistics, the frequency of dental caries has decreased in most industrialized nations over the past few decades. It has been suggested that it is due to the influence of multiple factors, including the use of fluoride, enhanced oral hygiene including brushing and flossing, dietary changes, and specific procedures performed in the dentist's office such as routine examinations, including diagnostic radiographs, scaling and polishing, fluoride applications, and sealants. Dental caries is a chronic, persistent dental condition that gets harder to cure as it progresses. The contemporary dental practice's preventive strategy has been acknowledged as a key factor in the recent drop in caries and a key component of the practice's service mix going forward. One of the World Health Organization's (WHO) major actions for ongoing oral health improvement is reorienting oral health services toward preventive and health promotion. A preventative approach can reduce the burden of oral health problems, as cited by WHO. Literature shows that although dentists' knowledge may be good, there are certain limitations to applying the preventive approach, lack of positive attitude, and implications in daily practice. With this background, the study aims to evaluate dental practitioners' knowledge, attitudes, and practice regarding caries preventive measures in Cairo compared to Riyadh.

ELIGIBILITY:
Inclusion Criteria:

* Licensed Egyptian and Saudi general dentists.

Exclusion Criteria:

* Undergraduate dental students
* Dental specialists
* Dentists who refused to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All Licenced General Dentisits from Cairo and Riyadah
Sampling Method: Non-Probability Sample
Enrollment: 248 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Knowledge, attitude and practice (KAP) of Dental Practitioners in Cairo and Riyadh | 1 year
  The study will be conducted via an online questionnaire
  The questionnaire is composed of the following sections:
  (A) Sociodemographic data including participants' age, gender, qualification, experience years, place of practice, and the number of pediatric patients seen every week.
  (B) Participants' knowledge of caries preventive measures. (C) Participants' attitudes and knowledge related to caries preventive measures.
  (D) Barriers in caries risk assessment and management practices.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

REFERENCES:
- [Background] Petersen PE. Priorities for research for oral health in the 21st century--the approach of the WHO Global Oral Health Programme. Community Dent Health. 2005 Jun;22(2):71-4. PMID 15984131
- [Background] Kitchens DH. The economics of pit and fissure sealants in preventive dentistry: a review. J Contemp Dent Pract. 2005 Aug 15;6(3):95-103. PMID 16127477
- [Background] Frame PS, Sawai R, Bowen WH, Meyerowitz C. Preventive dentistry: practitioners' recommendations for low-risk patients compared with scientific evidence and practice guidelines. Am J Prev Med. 2000 Feb;18(2):159-62. doi: 10.1016/s0749-3797(99)00138-5. PMID 10698247
- [Background] Farsi NM. The effect of education upon dentists' knowledge and attitude toward fissure sealants. Odontostomatol Trop. 1999 Jun;22(86):27-32. PMID 11372092
- [Background] Ghasemi H, Murtomaa H, Torabzadeh H, Vehkalahti MM. Knowledge of and Attitudes towards Preventive Dental Care among Iranian Dentists. Eur J Dent. 2007 Oct;1(4):222-9. PMID 19212471
- [Background] Patil RU, Sahu A, Kambalimath HV, Panchakshari BK, Jain M. Knowledge, Attitude and Practice among Dental Practitioners Pertaining to Preventive Measures in Paediatric Patients. J Clin Diagn Res. 2016 Dec;10(12):ZC71-ZC75. doi: 10.7860/JCDR/2016/22300.9122. Epub 2016 Dec 1. PMID 28209009